CLINICAL TRIAL: NCT00429910
Title: Chronic Myeloid Leukemia (CML) Cohort
Brief Title: Natural History Study of Patients With Chronic Myelogenous Leukemia
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jerome Ritz, MD, Jerome M.Ritz MD, Dana-Farber Cancer Institute
Other Study IDs: 03-015; P30CA006516 (NIH); CDR0000352370
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Leukemia
Keywords: accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Gathering information about patients with chronic myelogenous leukemia may help doctors learn more about the disease and find better methods of treatment and on-going care.

PURPOSE: This natural history study is collecting health information and disease-related information over time from patients with newly diagnosed chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the impact of current procedures for diagnosis, management, and follow-up on disease status of patients with newly diagnosed chronic myelogenous leukemia (CML).
* Determine the natural history of patients with CML who achieve response to imatinib mesylate.
* Determine the health perceptions, symptoms, insurance issues, and work issues of these patients.
* Determine whether medication compliance and planned dose reduction affect imatinib mesylate effectiveness in these patients.
* Determine the molecular and biologic factors associated with disease progression and good and poor response to imatinib mesylate in these patients.

OUTLINE: This is a longitudinal, prospective, cohort study.

Patients complete quality of life, functional status, medical and treatment history, and medication questionnaires at baseline and then every 6 months for 5 years.

Blood samples are collected at baseline and then every 6 months for 5 years. Specimens may be examined in the future in gene array studies and mutation analyses.

ELIGIBILITY:
Age 18 years and over Diagnosis within one year of enrollment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic myelogenous leukemia of any phase
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2003-02; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Impact of current procedures for diagnosis, management, and follow-up on disease status | 5 years
Natural history of patients with chronic myelogenous leukemia who achieve response to imatinib mesylate | 5 years
Health perceptions, symptoms, insurance issues, and work issues | 5 years
Affect of medication compliance and planned dose reduction on imatinib mesylate effectiveness | 5 years
Molecular and biologic factors associated with disease progression and good and poor response to imatinib mesylate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Ritz, MD, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No